CLINICAL TRIAL: NCT05430009
Title: Phase I Trial of Feasibility and Safety of Liver SBRT in Combination With Immune Checkpoint Inhibition in Patients With Metastatic Non-small Cell Lung Cancer
Brief Title: Liver SBRT in Combination With Immune Checkpoint Inhibition in Patients With Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Collaborators: LUNGevity Foundation (Other)
Responsible Party: Principal Investigator, Michael Green, Attending Physician, Radiation Oncology, VA Ann Arbor Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1652440
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Liver Metastases; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): This is an open-label, single-arm, single center clinical trial to evaluate the feasibility of liver SBRT (up to 4 metastases) during the first cycle of physician's choice ICI for NSCLC.
  Interventions: Radiation: Liver SBRT; Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Liver SBRT — 24-45 Gy delivered in 3-5 fractions to 1-4 lesions.
Drug: Pembrolizumab — 200 mg every 3 weeks or 400 mg every 6 weeks

SUMMARY:
Determine the feasibility of liver stereotactic body radiation therapy (SBRT) given in combination with systemic therapy (immune checkpoint inhibitors) in adult patients with metastatic NSCLC with liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age)
* Histologically or cytologically confirmed NSCLC with liver metastases
* Eligible for immune checkpoint inhibitors per treating medical oncologist
* Disease must be measurable per RECIST criteria
* ECOG Performance status of 0 - 2
* Adequate organ function per protocol.
* Allowable prior therapy includes adjuvant durvalumab, prior radiotherapy outside the upper abdomen.
* Patients must be willing and able to sign an informed consent form.
* Participants of childbearing potential willing to undergo pregnancy test and use contraception per Appendix.

Exclusion Criteria:

* Liver tumor burden which cannot be targeted with SBRT per treating radiation oncologist
* Presence of uncontrolled intercurrent illness or significant comorbidities precluding participation in a clinical study as determined by investigator
* Diagnosis of underlying parenchymal end stage liver disease (cirrhosis) or biliary disease (primary biliary cirrhosis).
* Other invasive malignancy active within 1 years, excluding in situ cancers
* Presence of psychiatric or substance abuse disorders that would interfere with compliance or safety
* Has a known history of active Bacillus Tuberculosis (TB), Hepatitis B or Hepatitis C infection
* Has received a live (active) vaccine within 30 days of enrollment.
* Active autoimmune disease that has required systemic treatment in the past 1 years aside from hormone replacement therapy (ie. thyroxine, insulin, or physiologic corticosteroid replacement therapy)
* Baseline corticosteroid use (>10 mg prednisone daily or equivalent) at study entry
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who receive all fractions of radiotherapy as planned | Up to 0.5 years after start of study treatment
  Feasibility determination. Analyzed with descriptive statistics.

SECONDARY OUTCOMES:
Proportion of patients who develop grade 3 or higher toxicity | Up to 1 year after start of study treatment
  Any serious adverse event that occurs within 60 days after treatment with SBRT or after this time frame and is considered related to the study treatment will also be reported. Analyzed with descriptive statistics.
Progression-free survival | Time Frame: Up to 3 years after end of study treatment
  PFS defined as the time from start of treatment to date of radiological or clinical progression (leading to withdrawal from the study), or death from any cause, whichever comes first. Assessed Per RECIST v1.1; analyzed using Kaplan-Meier curves and descriptive statistics.
Overall survival (OS) | Time Frame: Up to 3 years after end of study treatment
  OS defined as the time from start of treatment to death. This will be analyzed using Kaplan-Meier curves and descriptive statistics.
Proportion of patients with local control | Time Frame: Up to 3 years after end of study treatment
  Freedom from local progression (local control) is defined as the lack of progression of the tumors treated by RT, either by tumor size or enhancement. Progression or development of new tumors elsewhere in the liver or outside of the liver would not constitute a local control failure. Tumors which increase in size or demonstrate new or increasing enhancement are considered progression. Analyzed using Kaplan-Meier curves and descriptive statistics.

OTHER OUTCOMES:
Proportion of responders with increased frequency of circulating lymphocytes | Time Frame: Up to 3 years after end of study treatment
  Flow cytometry quantification of circulating biomarkers. Analyzed with paired T-test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Green, MD, Principal Investigator — VA Ann Arbor
Locations (1):
- Veterans Affairs Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No